CLINICAL TRIAL: NCT02375165
Title: Biomarkers for the Detection of Lymphatic Insufficiency
Acronym: Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine, Stanford University
Other Study IDs: 17690
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort with lymphedema: Participants with a history of acquired lymphedema of at least 6 months' duration, will have phlebotomy for serum and plasma.
  Interventions: Procedure: phlebotomy
- Cohort without lymphedema: Healthy volunteers; will have phlebotomy for serum and plasma.
  Interventions: Procedure: phlebotomy

INTERVENTIONS:
Procedure: phlebotomy — phlebotomy for collection of plasma and serum, ~30 cc
  Other Names: venipuncture

SUMMARY:
Acquired lymphedema is a disease that causes chronic swelling of the limb(s). It is frequently under-recognized or misdiagnosed. This study is designed to lead to the development of an accurate, noninvasive, blood test to allow testing for lymphedema. This approach is particularly useful to investigate relative responses to treatment interventions.

DETAILED DESCRIPTION:
The validation of a sensitive and specific biomarker assay for human acquired lymphatic vascular insufficiency would represent a highly significant development for the patient community. Accurate bioassay for the presence of lymphatic vascular insufficiency should help to pave the road for future human clinical trials of experimental drugs and therapies designed to treat human lymphatic diseases. Molecular profiling will be performed in human tissues (skin) obtained by biopsy. The insights gained from these initial analyses will determine the targets for assay in human body fluids (blood).

ELIGIBILITY:
Inclusion Criteria

For lymphedema participants:

* clinical diagnosis of lymphedema of at least 6 months' duration

Control participants:

* no evidence of lymphedema

Exclusion Criteria

For lymphedema participants:

* active cancer
* infection
* bleeding tendency
* active coronary artery disease
* congestive heart failure
* history of stroke or transient ischemic attack (TIA)
* uncontrolled hypertension
* renal insufficiency (serum creatinine > 1.1)
* active inflammatory or autoimmune disease (other than lymphedema)

For control participants:

* lymph node dissection
* radiation therapy
* active inflammatory disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive their care within Dr. Rockson's clinic in the Stanford Center for Lymphatic and Venous Disorders may be spoken to about voluntary participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-09; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers for the Detection of Lymphatic Vascular Insufficiency | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: Yes
to be determined
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available one year after the last study visit and for one year duration.
Access Criteria: Requestors will be required to complete a Data Access Agreement